CLINICAL TRIAL: NCT06106152
Title: A Single-center, Open Label, Exploratory Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of WTX212A Injection Combined With PD -1/PD-L1 Monoclonal Antibody in Patients With Advanced Lung Cancer
Brief Title: WTX212A Monotherapy and in Combination With PD -1/PD-L1 Monoclonal Antibody
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Westlake Therapeutics (Industry)
Responsible Party: Principal Investigator, Pingli Wang, Chief of Respiratory and Critical Care Medicine Department,pHD,MD, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Reboot-105
Record Dates: First submitted 2023-10-17; First posted 2023-10-30 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Advanced Lung Cancer

STUDY DESIGN:
Intervention Model Description: Single-center, open-label, exploratory study to evaluate the efficacy, safety, pharmacokinetics, and pharmacodynamics of WTX212A injection combined with PD -1/PD-L1 monoclonal antibody in patients with advanced lung cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fixed-dose in patients with advanced lung cancer (Experimental): WTX212A injection Fixed-dose in advanced lung cancer patients
  Interventions: Drug: WTX212A injection
- Combined Study in patients with advanced lung cancer (Experimental): Fixed-dose WTX212A injection combined with PD -1/PD-L1 monoclonal antibody in patients with advanced lung cancer
  Interventions: Drug: WTX212A injection; Drug: PD -1/PD-L1 monoclonal antibody

INTERVENTIONS:
Drug: WTX212A injection — The WTX212A infusion is given every 21 days
  Other Names: autologous red blood cell PD-1 inhibitor conjugate
Drug: PD -1/PD-L1 monoclonal antibody — The PD -1/PD-L1 monoclonal antibody is given every 21 days
  Other Names: PD -1/PD-L1antibody
  Arms: Combined Study in patients with advanced lung cancer

SUMMARY:
This trial is a single-center, open-label designed investigator-initiated clinical study (IIT) to evaluate the efficacy, safety, pharmacokinetics, and pharmacodynamics of WTX212A injection WTX212A injection combined with PD -1/PD-L1 monoclonal antibody in patients with advanced lung cancer

DETAILED DESCRIPTION:
The trial consist of Screening Period (30 days), Treatment Period (21*n days), Safety Follow-up Period (90 days) and Survival follow-up.

About 20 subjects are planned to be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* The subject signs an informed consent form, understands this study, is willing to follow and has the ability to complete all experimental procedures;
* Regardless of gender, aged 18 to 75 years old (including threshold);
* Histologically or cytologically confirmed locally advanced (stage IIB/IIC) or metastatic (stage IV) non-small cell lung cancer (NSCLC) with disease progression or intolerance after treatment or extensive stage small cell Lung cancer (SCLC)
* Patients with lung cancer who have been treated with at least 1 line system therapy or cannot currently receive standard therapy, and who have been treated with PD-1 or PD-L1 inhibitor antibody in the terminal line therapy regimen for ≥ 2 cycles;
* ECOG ≤1
* Expected life ≥ 3 months；
* Male participants, their spouses, and female participants of childbearing age should agree to use a medically recognized effective contraceptive method from the signing of the informed consent form until 3 months after the last administration;

Exclusion Criteria:

* People with other serious medical diseases, including but not limited to: uncontrolled diabetes, active peptic ulcer, active bleeding, etc., and people with uncontrollable or serious cardiovascular diseases,
* Patients with clinical symptoms and the need for repeated drainage of pleural and ascitic fluids;
* Previous or recent history of pulmonary fibrosis, severe lung function damage caused by pneumoconiosis, radiation pneumonia, and drug-related pneumonia;
* There have been adverse events related to the use of IO drugs that require permanent cessation of IO treatment;
* Known to have other malignant tumors, currently progressing or completing treatment at least once in the past 3 years. Exceptions include early tumors that have received radical treatment (carcinoma in situ or grade 1 tumor, non ulcerative primary melanoma with a depth of less than 1mm and no lymph nodes involved), skin basal cell carcinoma, skin squamous cell carcinoma, cervical carcinoma in situ, or breast carcinoma in situ that has received potential radical treatment;
* Subjects with symptomatic central nervous system (CNS) metastasis confirmed by imaging or pathological examination and clinically unstable for at least 14 days prior to enrollment who require steroid treatment;
* Having hereditary bleeding tendencies or coagulation disorders, or a history of thrombosis, hemolysis, or hemorrhagic diseases;
* Received significant surgical treatment or obvious traumatic injury within 28 days prior to the start of research treatment;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of WTX212A injection combined with PD -1/PD-L1 monoclonal antibody in the treatment of patients with IO- resistant advanced lung cancer. | 1 year
  Overall Response Rate (ORR) According to Response Evaluation Criteria In Solid Tumors Version 1.1

SECONDARY OUTCOMES:
the safety of WTX212A injection combined with PD -1/PD-L1 monoclonal antibody in the treatment of IO- resistant advanced lung cancer patients | 1 year
  The incidence of adverse events (AE), treatment related adverse events (TRAE), and severe adverse events (SAE) during the treatment of WTX212A injection
To evaluate the pharmacokinetic ( PK ) characteristics of WTX212A injection combined with PD -1/PD-L1 monoclonal antibody in patients with IO- resistant advanced lung cancer | 1 year
  Peak Plasma Concentration (Cmax)
To evaluate the immunogenicity of WTX212A injection combined with PD -1/PD-L1 monoclonal antibody in patients with IO -resistant advanced lung cancercheckpoint inhibitor resistance in advanced lung cancer patients | 1 year
  Describe the percentage of anti-drug antibodies (ADA) produced by subjects at each time point after treatment

OTHER OUTCOMES:
To evaluate the pharmacodynamics ( PD ) characteristics of WTX212A injection combined with PD -1/PD-L1 monoclonal antibody in patients with IO- resistant advanced lung cancer | 1 year
  The occupancy rate of PD-1 receptor on the surface of peripheral blood T cells in subjects after WTX212A infusion
To explore and evaluate WTX212A injection combined with PD -1/PD-L1 monoclonal antibody in the treatment of IO- resistant advanced lung cancer before and after treatment, analysis of immune cell subpopulations | 1 year
  Calculate the absolute values and percentages of immune cell subpopulations (absolute values and percentages of effector cells and immunosuppressive cells) before and after treatment of WTX212A injection combined with PD -1/PD-L1 monoclonal antibody in the treatment of IO -resistant advanced lung cancer. Immunomic analysis Variety
To explore and evaluate the changes in spleen size in patients with IO- resistant advanced lung cancer before and after treatment with WTX212A injection combined with PD -1/PD-L1 monoclonal antibody | 1 year
  Changes in spleen size before and after treatmen

CONTACTS AND LOCATIONS:
Overall Officials: pingli wang, phD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
There are no plans to disclose the data